CLINICAL TRIAL: NCT03651115
Title: Therapeutic Drug Monitoring of Gentamicin and Vancomycin, in Neonates, Using Dried Blood Spot Sampling.
Brief Title: TDM of Gentamicin and Vancomycin, in Neonates, Using Dried Blood Spot Sampling.
Acronym: MIDOMEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: MIDOMEN 16-024
Record Dates: First submitted 2018-08-13; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Blood Sample for Routine Care; Term or Premature Newborns (28 to 44 Amenorrhea Weeks); Gentamicin and/or Vancomycin
MeSH Terms: interventions — Drug Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonates with gentamicin
  Interventions: Diagnostic Test: therapeutic drug monitoring
- Neonates with vancomycin
  Interventions: Diagnostic Test: therapeutic drug monitoring

INTERVENTIONS:
Diagnostic Test: therapeutic drug monitoring — To monitor the blood concentrations of gentamicin and vancomycin

SUMMARY:
Gentamicin and vancomycin, widely used in neonatology, are antibiotics with a narrow therapeutic index and a risk of nephrotoxicity and ototoxicity. For these drugs, therapeutic drug monitoring (TDM) is required, to optimize the efficacy and tolerance of these antibiotics.

In newborns, the TDM of these antibiotics is really available, because of physiological features, such as renal elimination and hepatic metabolism which are both very dependent on age and maturation. Thus, in newborn, there is a large interindividual variability of pharmacokinetic parameters, making the dosage adjustment of antibiotics very difficult.

Unfortunately, because of a limited blood mass, the TDM of these antibiotics is very rarely practiced in these children. The introduction of a Died blood spot (DBS), which uses only a single drop of blood (<50 μL) preserved in dried form, thus makes it possible to reduce the blood volume taken and avoid the venous intrusion. The dosage needs the use of liquid chromatography coupled with tandem mass spectrometry (LC-MSMS), the only sensitive technique to work with such a low blood volume.

We therefore wish to develop this approach coupling DBS and LC-MSMS, in neonatology, to evaluate the concentration of these nephrotoxic antibiotics (gentamicin and vancomycin), as TDM. The blood concentrations of the antibiotic, per 100 new-born term or premature (50 gentamicin, 50 vancomycin), are compared to the physiological state of the child (premature or not, intrauterine growth retardation or not), its hemodynamic status (shock or not) and its efficacy / toxicity, evaluated by the clinician using a questionnaire.

The use of this new sampling method, as an alternative to conventional blood sampling, makes it possible to better monitor the concentrations of gentamicin and vancomycin in neonatalogy, thus reducing the risk of toxicity of these antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Term or premature newborns who receive one or two antibiotics (gentamicin, vancomycin) and who could benefit from pharmacological dosages of these drugs
* Premature from age 28 amenorrhea weeks
* Newborns up to 44 weeks corrected age
* Newborns at term / premature having a blood sample provided for routine care (capillary or venous sampling for blood glucose, blood gas, hemoglobinemia, sodium, potassium, lactate, bilirubin)

Exclusion Criteria:

* Premature before age 28 amenorrhea weeks corrected
* Newborns over 44 weeks of age corrected
* Hemostasis disorders
* Hemoglobinopathies
* Hearing or kidney malformation
* Absence of blood sampling as part of the routine care

Ages: 28 Weeks to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 new-born term or premature (50 gentamicin, 50 vancomycin)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Sampling time for vancomycin concentration | Day 3
Sampling time for gentamycin concentration | Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France